CLINICAL TRIAL: NCT00426101
Title: HLH-2004 Treatment Protocol
Brief Title: Treatment Protocol for Hemophagocytic Lymphohistiocytosis 2004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Meyer Children's Hospital IRCCS (Other); Leiden University Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); Ehime University Graduate School of Medicine (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Baylor College of Medicine (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); St. Anna Kinderkrebsforschung (Other); Hospital de Cruces (Other); Hospital JP Garrahan (Other Government)
Responsible Party: Principal Investigator, Jan-Inge Henter, Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLH-2004
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: Hemophagocytic lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Dexamethasone; Etoposide; Cyclosporine; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etoposide, Dexamethasone, Cyclosporin A plus IT MTX & Steroids (Experimental): As compared to the HLH-94 treatment, the main changes are that
  1. Cyclosporin A is administered from day 1 and
  2. Intrathecal steroids are added to the intrathecal methotrexate.
  Drugs, dosage, frequency and duration are described in the paragraph "Interventions" below.
  Interventions: Drug: Dexamethasone; Drug: Etoposide; Drug: Cyclosporin; Procedure: Intrathecal therapy; Procedure: Stem cell transplant

INTERVENTIONS:
Drug: Dexamethasone — 10 mg/m2 daily wk 1-2 5 mg/m2 daily wk 3-4 2.5 mg/m2 daily wk 5-6 1.25 mg/m2 daily wk 7 Steroids tapered wk 8
  If continuation:
  Pulses every 2nd wk, 10 mg/m2 for 3 days
Drug: Etoposide — 150 mg/m2 iv twice/wk (wk 1-2) 150 mg/m2 iv once/wk (wk 3-8)
  If continuation:
  150 mg/m2 iv, every 2nd wk
Drug: Cyclosporin — WK 1-8:
  - Aim at around 200 microgram/L (trough value). Start: 6 mg/kg daily (divided in 2 daily doses) wk 1, if kidney function is normal.
  If continuation:
  - Aim for around 200 microgram/L. Monitor GFR.
Procedure: Intrathecal therapy — If at 2 wks there are progressive neurological symptoms or if an abnormal CSF (cell count and protein) has not improved, then give 4 wkly intrathecal inj. Be aware that some pat may have increased intracranial pressure.
  Methotrexate: <1 yr 6 mg, 1-2 yrs 8 mg, 2-3 yrs 10 mg, >3 yrs 12 mg. Prednisolone: <1 yr 4 mg, 1-2 yrs 6 mg, 2-3 yrs 8 mg, >3 yrs 10 mg.
Procedure: Stem cell transplant — The SCT procedure is up to the treating physician. However, a suggested regimen is provided.

SUMMARY:
Without therapy HLH is often fatal, and often rapidly fatal. The treatment protocol HLH-94 has improved survival markedly as compared to the survival earlier. We now aim to improve survival further.

DETAILED DESCRIPTION:
The most dangerous period after HLH diagnosis is the first 2 months. In HLH-2004 we provide additional therapy during this period as compared to in HLH-94.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfil the diagnostic criteria of HLH.

Exclusion Criteria:

* Prior cytotoxic or cyclosporin treatment for HLH.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 368 (Actual)
Dates: Start 2004-01; Primary Completion 2011-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Survival | 1-year after diagnosis

SECONDARY OUTCOMES:
Late effects | 5-years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Inge Henter, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Childhood Cancer Research Unit, Karolinska Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Henter JI, Horne A, Arico M, Egeler RM, Filipovich AH, Imashuku S, Ladisch S, McClain K, Webb D, Winiarski J, Janka G. HLH-2004: Diagnostic and therapeutic guidelines for hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2007 Feb;48(2):124-31. doi: 10.1002/pbc.21039. PMID 16937360
- [Result] Bergsten E, Horne A, Arico M, Astigarraga I, Egeler RM, Filipovich AH, Ishii E, Janka G, Ladisch S, Lehmberg K, McClain KL, Minkov M, Montgomery S, Nanduri V, Rosso D, Henter JI. Confirmed efficacy of etoposide and dexamethasone in HLH treatment: long-term results of the cooperative HLH-2004 study. Blood. 2017 Dec 21;130(25):2728-2738. doi: 10.1182/blood-2017-06-788349. Epub 2017 Sep 21. PMID 28935695
- [Derived] Bergsten E, Horne A, Hed Myrberg I, Arico M, Astigarraga I, Ishii E, Janka G, Ladisch S, Lehmberg K, McClain KL, Minkov M, Nanduri V, Rosso DA, Sieni E, Winiarski J, Henter JI. Stem cell transplantation for children with hemophagocytic lymphohistiocytosis: results from the HLH-2004 study. Blood Adv. 2020 Aug 11;4(15):3754-3766. doi: 10.1182/bloodadvances.2020002101. PMID 32780845